CLINICAL TRIAL: NCT00667368
Title: Home Screening for Bacterial Vaginosis to Prevent STDs
Brief Title: Bacterial Vaginosis Home Screening to Prevent STDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-0131; HHSN272201300012I
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2015-08-20

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; children; chlamydia; gonorrhea; mentronidazole; vaginal; women
MeSH Terms: conditions — Vaginosis, Bacterial; Chlamydia Infections; Gonorrhea | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Bi-monthly testing for BV without treatment.
- Intervention (Experimental): Metronidazole 500mg twice daily for 7 days for Bacterial Vaginosis (BV) detection
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Bi-monthly testing and treatment for BV with Metronidazole if BV is detected; 500mg twice daily for 7 days.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether regular screening (every 2 months) and treatment for bacterial vaginosis (BV [infection of the vagina]) will reduce the number of incidences of chlamydia and gonorrhea (sexually transmitted diseases) over the course of a year. Chlamydial and gonococcal infections will be determined by vaginal swab testing at 4, 8, and 12 months after enrollment. Subjects will include 1500 women aged 15-25 years who have clinical evidence of BV, with no symptoms. Subjects will be randomly assigned to 1 of 2 possible study groups: the intervention group (treatment of BV) or the control group (no BV treatment). Every 2 months, subjects will complete a home self-testing kit for screening of BV using a swab. If BV is detected by self-test, the subjects in the interventional group will receive a 7 day course of the antibiotic metronidazole. Participants will be involved in study related procedures for up to 12 months.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is characterized by an imbalance in the normal vaginal bacterial flora. In the United States (US), BV is very common, and the most common cause of vaginitis, affecting approximately 1 in 10 sexually active young women. Because BV is so common, interventions targeting BV could have a tremendous public health impact. This is a phase III randomized controlled trial, in which the primary objective is to determine whether regular screening (every two months) and treatment for asymptomatic BV can reduce the one-year incidence of chlamydial and gonococcal infections, compared to a control group of women who receive regular monitoring (every two months) for BV but no treatment. The secondary study objective is to determine demographic and behavioral factors associated with the acquisition of BV, its persistence among women who are not treated for this condition, its spontaneous resolution, and its recurrence in women who are treated for this condition. This study protocol will enroll 1500 sexually active females, aged 15 - 25 years, from 6 US cities involved in the Sexually Transmitted Infections Clinical Trials Group network (Birmingham, Durham, Raleigh, Pittsburgh, Baltimore and San Francisco). To be eligible, women must have 2 or more risk factors for sexually transmitted diseases (STDs) and must have clinical evidence of asymptomatic BV at enrollment. For the purposes of this study, women with a vaginal pH>4.5 with >20 percent clue cells detected by microscopy to have asymptomatic BV. In addition, women must deny the presence of unusual or abnormal vaginal discharge or odor. Subjects will receive bi-monthly (every two months) home self-testing kits for BV using a vaginal swab. If BV is detected by self-test, the subjects in the intervention group will receive antibiotic treatment consisting of metronidazole 500mg twice daily for 7 days. Subjects will be randomized to either an intervention group (screening and treatment for BV) or a control group (monitoring for BV without treatment). Subjects in both the intervention group and the control group will complete bi-monthly (every 2 months) follow-up assessments for BV at months 2, 4, 6, 8, 10, and 12 (the final follow-up). In addition, subjects will provide sample collections for Chlamydia trachomatis and Neisseria gonorrhoeae at 4, 8, and 12 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

-Subject provides written informed consent, or if subject is under age 18, parent signs informed consent and subject signs assent. -Female age 15-25 years (age at last birthday). -Vaginal intercourse within the past 3 months. -Asymptomatic bacterial vaginosis (BV) a. Vaginal pH > 4.5 b. Clue cells on wet prep microscopy, >20 percent c. Woman denies unusual or abnormal vaginal odor and discharge. -Two or more risk factors for sexually transmitted diseases (STDs): a. Age less than or equal to 20 b. African-American race c. Hispanic ethnicity d. Regular douching (at least one time per month) e. Two or more sex partners (past 12 months) f. Current or past STD (past 12 months). -Be able to understand study procedures . -Be able to comply with the study procedures for the entire length of the study.

Exclusion Criteria:

-Self-reported pregnancy, or no menstrual period in past 4 weeks and positive urine pregnancy test Note: We will exclude women who are pregnant at the time of enrollment because some guidelines recommend screening and treatment for bacterial vaginosis (BV) in high-risk women during pregnancy. -Regular use of antibiotics: use at least once daily for 2 of the past six months ( e.g., for acne). Note: Women taking antibiotics on a regular basis will be excluded because antibiotic use could affect both BV and chlamydia/gonorrhea infections. -Self-reported currently married/partnered and living with husband/partner of over 1 year. This does not include married women who are separated. Note: We will exclude women who are married and who are in established long term relationships because our goal is to enroll a sample of women at high-risk for sexually transmitted diseases (STDs). Although these women are at risk for STDs, they are at lower risk overall than women who are single, separated, or divorced. -Homeless Note: We will exclude women who are homeless because they are likely to be difficult to track. -Excessive alcohol use (consumes more than 14 alcoholic drinks per week, or is not willing to abstain from alcohol for one week in order to take medication). Note: We will exclude persons who do not think they could avoid drinking alcohol for one week to take an antibiotic (because metronidazole plus alcohol can lead to nausea and vomiting). -Allergy to metronidazole. -Current or history of seizure disorder. -Current or history of any kind of neuropathy. -Use of warfarin sodium (Coumadin ®). -Use of cimetidine (Tagamet ®). -Known liver disease. Note: we will exclude women with current seizure disorders, women taking warfarin (Coumadin), women taking cimetidine, and women with known liver disease; as such women may be at greater risk of adverse consequences from taking metronidazole. -History of hysterectomy. Note: we will exclude women who have had a hysterectomy because most chlamydial and gonococcal infections target the cervix. -Trichomonas vaginalis detected via wet mount during eligibility assessment. Note: we will also exclude women with a trichomonas infection identified during eligibility assessment through wet mount evaluation because we will treat them with a single dose of metronidazole. Such treatment would affect BV among women in the study. Women treated with metronidazole during eligibility assessment will have to wait for one month post treatment to become eligible for the study. -Unable to swallow pills. -Has an active uncontrolled medical condition, such as cancer, or per the judgment of the principal investigator should not participate in the study. -Women who are in the menstrual phase of the menstrual cycle. -Current participation in another research study of an investigational drug. -For women younger than age 18 years (19 in Alabama), a parent or guardian they live with is unaware that she is sexually active.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1370 (Actual)
Dates: Start 2008-07-28 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - San Francisco Department of Public Health - San Francisco City Clinic, San Francisco, California
  - RTI International - Women's Global Health Imperative, San Francisco, California
  - Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland
  - University of North Carolina School of Medicine - Center for Infectious Diseases, Chapel Hill, North Carolina
  - Durham County Health Department, Durham, North Carolina
  - Magee Women's Hospital of UPMC - Reproductive Infectious Disease Research, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Schwebke JR, Lee JY, Lensing S, Philip SS, Wiesenfeld HC, Sena AC, Trainor N, Acevado N, Saylor L, Rompalo AM, Cook RL. Home Screening for Bacterial Vaginosis to Prevent Sexually Transmitted Diseases. Clin Infect Dis. 2016 Mar 1;62(5):531-6. doi: 10.1093/cid/civ975. Epub 2015 Nov 26. PMID 26611782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target enrollment was 1370 and 1370 participants were randomized, but 5 participants were later found to be enrolled twice. The second enrollment of these participants were removed; therefore, the total enrolled was 1365.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 682 | 683
Completed | 482 | 511
Not Completed | 200 | 172
Not completed — Lost to Follow-up | 176 | 155
Not completed — Discontinued early | 24 | 17

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 682 | 683 | 1365
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2) | 21 (2) | 21 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 682 | 683 | 1365
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 60 | 122
  Not Hispanic or Latino | 620 | 623 | 1243
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 11 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 9 | 4 | 13
  Black or African American | 535 | 530 | 1065
  White | 45 | 65 | 110
  More than one race | 54 | 48 | 102
  Unknown or Not Reported | 26 | 29 | 55
Region of Enrollment [Number; unit: participants]
  United States | 682 | 683 | 1365

OUTCOME MEASURES:

1. Primary Outcome: One-year Incidence of Chlamydial and Gonococcal Infections in Women Who Receive Screening (Every 2 Months) and Treatment for Asymptomatic Bacterial Vaginosis as Compared to a Control Group With Regular Monitoring (Every 2 Months) But no Treatment
Description: Chlamydia and gonococcal infections were determined by vaginal swab testing collected at 4, 8, and 12 months after enrollment. Specimens were evaluated using the BD ProbeTec Amplified DNA AssayTM (Becton-Dickson, Inc. Sparks, MD). The primary outcome measure is the combined number of chlamydia and gonococcal infections.
Time Frame: At 4, 8, and 12 months after enrollment.
Measure: Number (95% Confidence Interval); unit: Number infections per 100 person-years
Arm/Group | Control | Intervention
Number analyzed (Participants) | 682 | 683
Number infections per 100 person-years | 19.2 [15.9 to 23.2] | 18.3 [15.1 to 22.1]
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.754, Two-sample test, Poisson; Risk Difference (RD) = -0.9, 95% CI 2-sided [-12.0 to 10.1] — The risk difference reflects the treatment arm minus the control arm. The units are the number of positive tests for chlamydia and gonorrhea per 100 person-years

2. Secondary Outcome: Percentage of Women Testing Positive for Bacterial Vaginosis (BV) Through 12 Months
Description: Percentage of women testing positive for BV at any follow-up visit. The outcome of BV status was determined by self-collected vaginal swab specimens that were evaluated by the Nugent criteria. A Nugent score of 7-10 indicates positive for BV.
Time Frame: 2, 4, 6, 8, 10, 12 months after enrollment
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 682 | 683
percentage of participants | 92.5 | 82.6
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 12 months after enrollment
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 3/682 | 7/683
Other Adverse Events (participants affected / at risk) | 0/682 | 0/683
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=682) | Intervention (N=683)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral Disk Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Turbo-Ovarian Abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1)
Optic Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Postpartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No